CLINICAL TRIAL: NCT04818996
Title: Evaluation of the Effect of Mediterranean Diet on Body Composition, Oxidant Stress and Proinflammatory Markers in Breast Cancer Patients
Brief Title: Evaluation of the Effect of Mediterranean Diet on Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Burcu Deniz Gunes, Research Assistant, Aydin Adnan Menderes University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019/044
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer
Keywords: Diet therapy; Mediterranean diet; Oxidant Stress markers; Proinflammatory markers; Body Composition
MeSH Terms: conditions — Breast Neoplasms | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mediterranean Diet (Experimental): In the study, the participants were applied a diet compatible with the Mediterranean diet for 8 weeks.
  Interventions: Behavioral: Mediterranean Diet

INTERVENTIONS:
Behavioral: Mediterranean Diet — While calculating the energy of the Mediterranean diet applied to the individuals participating in the study, Mifflin-St. Jeor equation is used. The macronutrient composition of the Mediterranean diet was calculated as 36-40% fat, 40-45% carbohydrate and 15-20% protein. This diet is enriched with natural foods (fruits, vegetables, legumes, whole grain foods, fish, olive oil and oilseeds such as walnuts and almonds).
  In addition, anthropometric measurements and body composition analysis of the participants were performed both at the beginning and at the end of the study, and some biochemical parameters (IL-6, TNF-α, CRP, MDA, TAS, TOS and routine blood parameters) were evaluated.

SUMMARY:
In this study, it was aimed to evaluate the effect of the Mediterranean diet on body composition, oxidant stress and proinflammatory markers in overweight and obese breast cancer women.

DETAILED DESCRIPTION:
Breast cancer is the most common type of cancer among women in both developed and developing countries and is the leading cause of cancer death among women worldwide. Breast cancer is a disease that can develop and progress for various reasons. In addition to unchangeable factors such as increasing age and genotype, modifiable factors such as smoking, alcohol consumption, lack of physical activity, malnutrition, and obesity play a role in the pathogenesis of the disease.

Breast cancer risk increases with increasing body mass index (BMI) in postmenopausal women. Chronic inflammation in obesity is associated with an increase in the release of proinflammatory factors (such as TNF-α, IL-1, IL-6). This situation; It is a risk factor for many types of cancer such as colon, stomach, breast and prostate carcinomas and supports a cause-effect relationship between obesity and cancer. These proinflammatory factors act as signal converters for tumor growth and progression. Obese women have elevated levels of TNF-α and IL-6 in the circulation, and this is associated with the development and progression of breast tumors.

The Mediterranean Diet, which consists of high amounts of monounsaturated fatty acids, fruits, vegetables and whole grains, has been widely evaluated and indicated as an important factor in preventing tumor formation from inflammatory pathways.

Weight loss improves the antitumor immune system, lowers estrogen levels, reduces the risk of breast cancer and has been associated with better outcomes in obese patients. Lifestyle intervention studies strongly suggest that weight loss is possible and observational studies can actually improve breast cancer survival.In this regard, a healthy lifestyle and diet are the first steps to prevent breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old,
* BMI value to be ≥25 kg/m2,
* To be diagnosed with breast cancer stage I, II or III,
* Being a positive hormone receptor status, one of the biological subtypes of breast cancer,
* Having completed chemotherapy and / or radiotherapy treatment at least 6 months before starting the study,
* Not applying any treatment for body weight loss,
* Accepting to participate in the study,
* Perceiving disorder and not having communication problems.

Exclusion Criteria:

* Being under the age of 18 and over the age of 65,
* BMI value to be 40 kg/m2,
* Having advanced stage breast cancer (IV and V),
* Being diagnosed with cancer or metastasis in other organs,
* Being one of the biological subtypes of breast cancer, hormone receptor status being negative,
* Using antioxidant vitamin-mineral supplements,
* Using herbal supplements,
* Being pregnant or planning a pregnancy,
* To stop working after starting diet therapy.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with breast cancer
Enrollment: 25 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline, 8 weeks
  Body weight (kg) was measured using the InBody 270 brand device.
Change in body mass indexs | Baseline, 8 weeks
  The BMI is defined as the body mass divided by the square of the body height, and is expressed in units of kg/m^2, resulting from mass in kilograms and height in metres.
Change in fat mass measured by bioelectrical impedance analyzer | Baseline, 8 weeks
  Fat mass (kg) was measured using the InBody 270 brand device.
Change in fat-free mass measured by bioelectrical impedance analyzer | Baseline, 8 weeks
  Fat-free mass (kg) was measured using the InBody 270 brand device.
Change in resting metabolic rate (RMR) measured by bioelectrical impedance analyzer | Baseline, 8 weeks
  RMR (kcal) was measured using the InBody 270 brand device.
Change in interleukin 6 (IL-6) | Baseline, 8 weeks
  Blood was drawn from participants for assessment of IL-6 (pg/mL) at the beginning and end of the study after fasting for at least 8 hours
Change in tumor necrosis factor alpha (TNF-α) | Baseline, 8 weeks
  Blood was drawn from participants for assessment of TNF-α (pg/mL) at the beginning and end of the study after fasting for at least 8 hours
Change in malondialdehyde (MDA) | Baseline, 8 weeks
  Blood was drawn from participants for assessment of MDA (mmol/L) at the beginning and end of the study after fasting for at least 8 hours
Change in total antioxidant status (TAS) | Baseline, 8 weeks
  Blood was drawn from participants for assessment of TAS (mmol/L) at the beginning and end of the study after fasting for at least 8 hours
Change in total oxidant status (TOS) | Baseline, 8 weeks
  Blood was drawn from participants for assessment of TOS (µmol/L) at the beginning and end of the study after fasting for at least 8 hours

SECONDARY OUTCOMES:
Change in waist circumference | Baseline, 8 weeks
  Waist circumference (cm) was measured with a non-stretch tape measure.
Change in hip circumference | Baseline, 8 weeks
  Hip circumference (cm) was measured with a non-stretch tape measure.
Change in dietary inflammatory index (DII) | Baseline, 8 weeks
  Dietary inflammatory index (DII) was calculated with 3-day food consumption record.
Change in oxidative stress index (OSI) | Baseline, 8 weeks
  The oxidative stress index (OSI) value expressed as a percentage of the ratio of serum total oxidant status (TOS) levels to total antioxidant status (TAS) levels was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu Deniz Güneş, Study Chair — Aydın Adnan Menderes University, Faculty of Health Sciences, Department of Nutrition and Dietetics
Locations (1):
- Aydın Adnan Menderes University, Faculty of Health Sciences, Department of Nutrition and Dietetics, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.